CLINICAL TRIAL: NCT02045290
Title: Metformin Therapy for Overweight Adolescents With Type 1 Diabetes (T1D)--Insulin Clamp Ancillary Study for Assessment of Insulin Resistance
Brief Title: Insulin Clamp Ancillary Study for Assessment of Insulin Resistance
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: T1DX Insulin Clamp Ancillary
Record Dates: First submitted 2014-01-15; First posted 2014-01-24 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2017-03

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oral Placebo (Placebo Comparator): A central pharmacy will compound a placebo to match the metformin tablets.
  The placebo product will contain the following components:
  * Micosolle™, silica based excipient
  * Silicified Micro Crystalline Cellulose, National Formulary
  * Safflower Oil, United States Pharmacopeia
  * K-30 Povidone Powder
  * Magnesium Stearate, National Formulary (Vegetable source)
  * Fumed Silica, National Formulary
  Interventions: Drug: Placebo
- Metformin (Experimental): Metformin 2000 mg per day
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — The strength of each tablet will be 500 mg. Participants will build up to a daily dose over four weeks by taking one tablet per day for 7 days, one tablet twice daily for 7 days, one tablet in the morning and 2 tablets at night for 7 days, and then 2 tablets in the morning and 2 tablets at night, daily throughout the remainder of the study treatment period.
  Arms: Metformin
Drug: Placebo
  Arms: Oral Placebo

SUMMARY:
Insulin Clamp Ancillary study for Assessment of Insulin Resistance will be conducted as a sub-study to the main protocol, Metformin Therapy for Overweight Adolescents With Type 1 Diabetes (NCT01881828). The purpose of this ancillary study is to assess if metformin will improve tissue-specific insulin resistance (IR) in type 1 diabetes using a hyperinsulinemic euglycemic clamp; a 3-month randomized trial comparing metformin versus placebo in 12 to <20 year olds with BMI >85th percentile ( total daily insulin dose >0.7 units/kg, and HbA1c 7.0%-9.9%).

ELIGIBILITY:
Inclusion Criteria:

1. Meets eligibility criteria of the main study, Metformin Therapy for Overweight Adolescents With Type 1 Diabetes (NCT01881828).

Exclusion Criteria:

1. Low hemoglobin or hematocrit as defined by each local institution's rules for insulin clamps or if no institutional requirements a Hematocrit <30% or hemoglobin <10 gm/dL

Ages: 12 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 37 (Actual)
Dates: Start 2014-01; Primary Completion 2016-02-15 (Actual); Study Completion 2016-02-15 (Actual)

PRIMARY OUTCOMES:
Change in insulin resistance (IR) from baseline to 13 weeks | 0-13 weeks
  Hyperinsulinemic euglycemic clamp to assess metformin's impact on muscle IR via glucose infusion rate (GIR).

SECONDARY OUTCOMES:
Change in Hepatic IR from baseline to 13 weeks | 0-13 weeks
  Graded hyperinsulinemic euglycemic clamp with glucose and glycerol isotopes to assess metformin's impact on:
  • Hepatic IR
Change in Adipose IR from baseline to 13 weeks | 0-13 weeks
  Graded hyperinsulinemic euglycemic clamp with glucose and glycerol isotopes to assess metformin's impact on:
  • Adipose IR

CONTACTS AND LOCATIONS:
Overall Officials: Kellee M Miller, MPH, Principal Investigator — Jaeb Center for Health Research; Ingrid Libman, MD, PhD, Study Chair — Childrens Hospital of University of Pittsburgh Medical Center; Kristen Nadeau, MD, Study Chair — University of Colorado Denver/Childrens Hospital Colorado
Locations (1):
- Jaeb Center for Health Research, Tampa, Florida, United States

REFERENCES:
- [Background] Snell-Bergeon JK, Hokanson JE, Jensen L, MacKenzie T, Kinney G, Dabelea D, Eckel RH, Ehrlich J, Garg S, Rewers M. Progression of coronary artery calcification in type 1 diabetes: the importance of glycemic control. Diabetes Care. 2003 Oct;26(10):2923-8. doi: 10.2337/diacare.26.10.2923. PMID 14514603
- [Background] Maahs DM, Kinney GL, Wadwa P, Snell-Bergeon JK, Dabelea D, Hokanson J, Ehrlich J, Garg S, Eckel RH, Rewers MJ. Hypertension prevalence, awareness, treatment, and control in an adult type 1 diabetes population and a comparable general population. Diabetes Care. 2005 Feb;28(2):301-6. doi: 10.2337/diacare.28.2.301. PMID 15677783
- [Background] Wadwa RP, Kinney GL, Maahs DM, Snell-Bergeon J, Hokanson JE, Garg SK, Eckel RH, Rewers M. Awareness and treatment of dyslipidemia in young adults with type 1 diabetes. Diabetes Care. 2005 May;28(5):1051-6. doi: 10.2337/diacare.28.5.1051. PMID 15855566
- [Background] Borch-Johnsen K, Kreiner S. Proteinuria: value as predictor of cardiovascular mortality in insulin dependent diabetes mellitus. Br Med J (Clin Res Ed). 1987 Jun 27;294(6588):1651-4. doi: 10.1136/bmj.294.6588.1651. PMID 3113569
- [Background] Krolewski AS, Kosinski EJ, Warram JH, Leland OS, Busick EJ, Asmal AC, Rand LI, Christlieb AR, Bradley RF, Kahn CR. Magnitude and determinants of coronary artery disease in juvenile-onset, insulin-dependent diabetes mellitus. Am J Cardiol. 1987 Apr 1;59(8):750-5. doi: 10.1016/0002-9149(87)91086-1. PMID 3825934
- [Background] Snell-Bergeon JK, Hokanson JE, Kinney GL, Dabelea D, Ehrlich J, Eckel RH, Ogden L, Rewers M. Measurement of abdominal fat by CT compared to waist circumference and BMI in explaining the presence of coronary calcium. Int J Obes Relat Metab Disord. 2004 Dec;28(12):1594-9. doi: 10.1038/sj.ijo.0802796. PMID 15467773
- [Background] Maahs DM, Ogden LG, Kinney GL, Wadwa P, Snell-Bergeon JK, Dabelea D, Hokanson JE, Ehrlich J, Eckel RH, Rewers M. Low plasma adiponectin levels predict progression of coronary artery calcification. Circulation. 2005 Feb 15;111(6):747-53. doi: 10.1161/01.CIR.0000155251.03724.A5. Epub 2005 Feb 7. PMID 15699257
- [Background] Orchard TJ, Olson JC, Erbey JR, Williams K, Forrest KY, Smithline Kinder L, Ellis D, Becker DJ. Insulin resistance-related factors, but not glycemia, predict coronary artery disease in type 1 diabetes: 10-year follow-up data from the Pittsburgh Epidemiology of Diabetes Complications Study. Diabetes Care. 2003 May;26(5):1374-9. doi: 10.2337/diacare.26.5.1374. PMID 12716791
- [Background] Libby P, Nathan DM, Abraham K, Brunzell JD, Fradkin JE, Haffner SM, Hsueh W, Rewers M, Roberts BT, Savage PJ, Skarlatos S, Wassef M, Rabadan-Diehl C; National Heart, Lung, and Blood Institute; National Institute of Diabetes and Digestive and Kidney Diseases Working Group on Cardiovascular Complications of Type 1 Diabetes Mellitus. Report of the National Heart, Lung, and Blood Institute-National Institute of Diabetes and Digestive and Kidney Diseases Working Group on Cardiovascular Complications of Type 1 Diabetes Mellitus. Circulation. 2005 Jun 28;111(25):3489-93. doi: 10.1161/CIRCULATIONAHA.104.529651. No abstract available. PMID 15983263
- [Background] Lloyd CE, Kuller LH, Ellis D, Becker DJ, Wing RR, Orchard TJ. Coronary artery disease in IDDM. Gender differences in risk factors but not risk. Arterioscler Thromb Vasc Biol. 1996 Jun;16(6):720-6. doi: 10.1161/01.atv.16.6.720. PMID 8640398
- [Background] Soedamah-Muthu SS, Chaturvedi N, Toeller M, Ferriss B, Reboldi P, Michel G, Manes C, Fuller JH; EURODIAB Prospective Complications Study Group. Risk factors for coronary heart disease in type 1 diabetic patients in Europe: the EURODIAB Prospective Complications Study. Diabetes Care. 2004 Feb;27(2):530-7. doi: 10.2337/diacare.27.2.530. PMID 14747240
- [Background] Amiel SA, Sherwin RS, Simonson DC, Lauritano AA, Tamborlane WV. Impaired insulin action in puberty. A contributing factor to poor glycemic control in adolescents with diabetes. N Engl J Med. 1986 Jul 24;315(4):215-9. doi: 10.1056/NEJM198607243150402. PMID 3523245
- [Background] Arslanian S, Heil BV, Kalhan SC. Hepatic insulin action in adolescents with insulin-dependent diabetes mellitus: relationship with long-term glycemic control. Metabolism. 1993 Mar;42(3):283-90. doi: 10.1016/0026-0495(93)90075-y. PMID 8487645
- [Background] Arslanian S, Nixon PA, Becker D, Drash AL. Impact of physical fitness and glycemic control on in vivo insulin action in adolescents with IDDM. Diabetes Care. 1990 Jan;13(1):9-15. doi: 10.2337/diacare.13.1.9. PMID 2404722
- [Background] Heptulla RA, Stewart A, Enocksson S, Rife F, Ma TY, Sherwin RS, Tamborlane WV, Caprio S. In situ evidence that peripheral insulin resistance in adolescents with poorly controlled type 1 diabetes is associated with impaired suppression of lipolysis: a microdialysis study. Pediatr Res. 2003 May;53(5):830-5. doi: 10.1203/01.PDR.0000059552.08913.B7. PMID 12702748
- [Background] Nadeau KJ, Regensteiner JG, Bauer TA, Brown MS, Dorosz JL, Hull A, Zeitler P, Draznin B, Reusch JE. Insulin resistance in adolescents with type 1 diabetes and its relationship to cardiovascular function. J Clin Endocrinol Metab. 2010 Feb;95(2):513-21. doi: 10.1210/jc.2009-1756. Epub 2009 Nov 13. PMID 19915016
- [Background] Purnell JQ, Hokanson JE, Marcovina SM, Steffes MW, Cleary PA, Brunzell JD. Effect of excessive weight gain with intensive therapy of type 1 diabetes on lipid levels and blood pressure: results from the DCCT. Diabetes Control and Complications Trial. JAMA. 1998 Jul 8;280(2):140-6. doi: 10.1001/jama.280.2.140. PMID 9669786
- [Background] Regensteiner JG. Type 2 diabetes mellitus and cardiovascular exercise performance. Rev Endocr Metab Disord. 2004 Aug;5(3):269-76. doi: 10.1023/B:REMD.0000032416.13070.01. No abstract available. PMID 15211099
- [Background] Regensteiner JG, Bauer TA, Reusch JE, Brandenburg SL, Sippel JM, Vogelsong AM, Smith S, Wolfel EE, Eckel RH, Hiatt WR. Abnormal oxygen uptake kinetic responses in women with type II diabetes mellitus. J Appl Physiol (1985). 1998 Jul;85(1):310-7. doi: 10.1152/jappl.1998.85.1.310. PMID 9655791
- [Background] Regensteiner JG, Bauer TA, Reusch JE, Quaife RA, Chen MY, Smith SC, Miller TM, Groves BM, Wolfel EE. Cardiac dysfunction during exercise in uncomplicated type 2 diabetes. Med Sci Sports Exerc. 2009 May;41(5):977-84. doi: 10.1249/MSS.0b013e3181942051. PMID 19346991
- [Background] Rewers M, Zaccaro D, D'Agostino R, Haffner S, Saad MF, Selby JV, Bergman R, Savage P; Insulin Resistance Atherosclerosis Study Investigators. Insulin sensitivity, insulinemia, and coronary artery disease: the Insulin Resistance Atherosclerosis Study. Diabetes Care. 2004 Mar;27(3):781-7. doi: 10.2337/diacare.27.3.781. PMID 14988302
- [Background] Haffner SM, D'Agostino R Jr, Mykkanen L, Tracy R, Howard B, Rewers M, Selby J, Savage PJ, Saad MF. Insulin sensitivity in subjects with type 2 diabetes. Relationship to cardiovascular risk factors: the Insulin Resistance Atherosclerosis Study. Diabetes Care. 1999 Apr;22(4):562-8. doi: 10.2337/diacare.22.4.562. PMID 10189532
- [Background] Nadeau KJ, Zeitler PS, Bauer TA, Brown MS, Dorosz JL, Draznin B, Reusch JE, Regensteiner JG. Insulin resistance in adolescents with type 2 diabetes is associated with impaired exercise capacity. J Clin Endocrinol Metab. 2009 Oct;94(10):3687-95. doi: 10.1210/jc.2008-2844. Epub 2009 Jul 7. PMID 19584191
- [Background] Perseghin G, Lattuada G, Danna M, Sereni LP, Maffi P, De Cobelli F, Battezzati A, Secchi A, Del Maschio A, Luzi L. Insulin resistance, intramyocellular lipid content, and plasma adiponectin in patients with type 1 diabetes. Am J Physiol Endocrinol Metab. 2003 Dec;285(6):E1174-81. doi: 10.1152/ajpendo.00279.2003. Epub 2003 Aug 21. PMID 12933352
- [Background] Greenfield JR, Samaras K, Chisholm DJ. Insulin resistance, intra-abdominal fat, cardiovascular risk factors, and androgens in healthy young women with type 1 diabetes mellitus. J Clin Endocrinol Metab. 2002 Mar;87(3):1036-40. doi: 10.1210/jcem.87.3.8324. PMID 11889158
- [Background] Taskinen MR. Quantitative and qualitative lipoprotein abnormalities in diabetes mellitus. Diabetes. 1992 Oct;41 Suppl 2:12-7. doi: 10.2337/diab.41.2.s12. PMID 1526330
- [Background] Nijs HG, Radder JK, Frolich M, Krans HM. The course and determinants of insulin action in type 1 (insulin-dependent) diabetes mellitus. Diabetologia. 1989 Jan;32(1):20-7. doi: 10.1007/BF00265399. PMID 2651185
- [Background] Yang X, Ongusaha PP, Miles PD, Havstad JC, Zhang F, So WV, Kudlow JE, Michell RH, Olefsky JM, Field SJ, Evans RM. Phosphoinositide signalling links O-GlcNAc transferase to insulin resistance. Nature. 2008 Feb 21;451(7181):964-9. doi: 10.1038/nature06668. PMID 18288188
- [Background] Dentin R, Hedrick S, Xie J, Yates J 3rd, Montminy M. Hepatic glucose sensing via the CREB coactivator CRTC2. Science. 2008 Mar 7;319(5868):1402-5. doi: 10.1126/science.1151363. PMID 18323454
- [Background] Koivisto VA, Yki-Jarvinen H. Changes in muscle glucose metabolism in type 1 diabetes. Ann Med. 1990 Jun;22(3):201-5. doi: 10.3109/07853899009147270. PMID 2393555
- [Background] Chibalin AV, Leng Y, Vieira E, Krook A, Bjornholm M, Long YC, Kotova O, Zhong Z, Sakane F, Steiler T, Nylen C, Wang J, Laakso M, Topham MK, Gilbert M, Wallberg-Henriksson H, Zierath JR. Downregulation of diacylglycerol kinase delta contributes to hyperglycemia-induced insulin resistance. Cell. 2008 Feb 8;132(3):375-86. doi: 10.1016/j.cell.2007.12.035. PMID 18267070
- [Background] Jensen MD, Caruso M, Heiling V, Miles JM. Insulin regulation of lipolysis in nondiabetic and IDDM subjects. Diabetes. 1989 Dec;38(12):1595-601. doi: 10.2337/diab.38.12.1595. PMID 2573554
- [Background] Nadeau KJ, Ehlers LB, Zeitler PS, Love-Osborne K. Treatment of non-alcoholic fatty liver disease with metformin versus lifestyle intervention in insulin-resistant adolescents. Pediatr Diabetes. 2009 Feb;10(1):5-13. doi: 10.1111/j.1399-5448.2008.00450.x. Epub 2008 Aug 20. PMID 18721166
- [Background] Moreau KL, Donato AJ, Seals DR, DeSouza CA, Tanaka H. Regular exercise, hormone replacement therapy and the age-related decline in carotid arterial compliance in healthy women. Cardiovasc Res. 2003 Mar;57(3):861-8. doi: 10.1016/s0008-6363(02)00777-0. PMID 12618248
- [Background] Ekstrand AV, Groop PH, Gronhagen-Riska C. Insulin resistance precedes microalbuminuria in patients with insulin-dependent diabetes mellitus. Nephrol Dial Transplant. 1998 Dec;13(12):3079-83. doi: 10.1093/ndt/13.12.3079. PMID 9870469
- [Background] DeFronzo RA, Simonson D, Ferrannini E. Hepatic and peripheral insulin resistance: a common feature of type 2 (non-insulin-dependent) and type 1 (insulin-dependent) diabetes mellitus. Diabetologia. 1982 Oct;23(4):313-9. doi: 10.1007/BF00253736. PMID 6754515
- [Background] Van Pelt RE, Gozansky WS, Hickner RC, Schwartz RS, Kohrt WM. Acute modulation of adipose tissue lipolysis by intravenous estrogens. Obesity (Silver Spring). 2006 Dec;14(12):2163-72. doi: 10.1038/oby.2006.253. PMID 17189542
- [Background] Druet C, Tubiana-Rufi N, Chevenne D, Rigal O, Polak M, Levy-Marchal C. Characterization of insulin secretion and resistance in type 2 diabetes of adolescents. J Clin Endocrinol Metab. 2006 Feb;91(2):401-4. doi: 10.1210/jc.2005-1672. Epub 2005 Nov 15. PMID 16291705
- [Background] Gilker CD, Pesola GR, Matthews DE. A mass spectrometric method for measuring glycerol levels and enrichments in plasma using 13C and 2H stable isotopic tracers. Anal Biochem. 1992 Aug 15;205(1):172-8. doi: 10.1016/0003-2697(92)90595-x. PMID 1443555
- [Background] STEELE R. Influences of glucose loading and of injected insulin on hepatic glucose output. Ann N Y Acad Sci. 1959 Sep 25;82:420-30. doi: 10.1111/j.1749-6632.1959.tb44923.x. No abstract available. PMID 13833973
- [Background] Finegood DT, Bergman RN, Vranic M. Estimation of endogenous glucose production during hyperinsulinemic-euglycemic glucose clamps. Comparison of unlabeled and labeled exogenous glucose infusates. Diabetes. 1987 Aug;36(8):914-24. doi: 10.2337/diab.36.8.914. PMID 3297886
- [Background] Kamel EG, McNeill G, Han TS, Smith FW, Avenell A, Davidson L, Tothill P. Measurement of abdominal fat by magnetic resonance imaging, dual-energy X-ray absorptiometry and anthropometry in non-obese men and women. Int J Obes Relat Metab Disord. 1999 Jul;23(7):686-92. doi: 10.1038/sj.ijo.0800904. PMID 10454101
- [Background] Sarnblad S, Kroon M, Aman J. Metformin as additional therapy in adolescents with poorly controlled type 1 diabetes: randomised placebo-controlled trial with aspects on insulin sensitivity. Eur J Endocrinol. 2003 Oct;149(4):323-9. doi: 10.1530/eje.0.1490323. PMID 14514347
- [Background] Martin FI, Hopper JL. The relationship of acute insulin sensitivity to the progression of vascular disease in long-term type 1 (insulin-dependent) diabetes mellitus. Diabetologia. 1987 Mar;30(3):149-53. doi: 10.1007/BF00274219. PMID 3556289
- [Background] Regensteiner JG, Sippel J, McFarling ET, Wolfel EE, Hiatt WR. Effects of non-insulin-dependent diabetes on oxygen consumption during treadmill exercise. Med Sci Sports Exerc. 1995 Jun;27(6):875-81. PMID 7658949
- [Derived] Cree-Green M, Bergman BC, Cengiz E, Fox LA, Hannon TS, Miller K, Nathan B, Pyle L, Kahn D, Tansey M, Tichy E, Tsalikian E, Libman I, Nadeau KJ. Metformin Improves Peripheral Insulin Sensitivity in Youth With Type 1 Diabetes. J Clin Endocrinol Metab. 2019 Aug 1;104(8):3265-3278. doi: 10.1210/jc.2019-00129. PMID 30938764